CLINICAL TRIAL: NCT05816382
Title: A Long-term Extension Study to Evaluate the Safety and Tolerability of TAK-861 in Participants With Selected Central Hypersomnia Conditions
Brief Title: A Study of TAK-861 for the Treatment of Selected Central Hypersomnia Conditions
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TAK-861-2003; U1111-1283-1888 (Other: WHO); jRCT2031230135 (Registry Identifier: jRCT); 2023-508462-15 (Other: EU CTIS)
Record Dates: First submitted 2023-03-31; First posted 2023-04-18 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Narcolepsy Type 1
Keywords: Drug Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TAK-861 Dose 1 (Experimental): Participants will receive TAK-861 dose 1 for up to approximately 5 years.
  Interventions: Drug: TAK-861
- TAK-861 Dose 2 (Experimental): Participants will receive TAK-861 dose 2 for up to approximately 5 years.
  Interventions: Drug: TAK-861

INTERVENTIONS:
Drug: TAK-861 — TAK-861 tablets

SUMMARY:
The main aim is to evaluate the safety and tolerability of TAK-861 on participants with type 1 narcolepsy, who were exposed to previously tested doses of TAK-861.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-861. TAK-861 is being tested to treat people who have narcolepsy type 1 (NT1). This study will look at the safety of TAK-861 along with improvement in narcolepsy symptoms, including excessive daytime sleepiness (EDS) and number of cataplexy episodes.

This study was initiated in parallel with the parent phase 2 studies, TAK-861-2001 (NCT05687903) and TAK-861-2002 (NCT05687916), which included participants with NT1 and narcolepsy type 2 (NT2), respectively. This long-term extension (LTE) study enrolled participants with both diagnoses from the two phase 2 studies. As the TAK-861-2002 study did not meet prespecified criteria, all participants with NT2 have been discontinued, and this extension study will only include participants with NT1 who previously completed a parent study. Additional parent studies include all TAK-861 phase 3 studies.

The study will enroll up to 500 patients. Participants will be assigned to one of the treatment groups according to the dose assigned to them in their parent study. Similarly, participants who were previously on a placebo dose will also be assigned to one of the treatment groups randomly. All participants in the study will receive TAK-861.

Participants with NT1 will receive the following dose from the parent study:

* TAK-861 Dose 1
* TAK-861 Dose 2

This multi-center trial will be conducted worldwide. The overall time to participate in this study is up to approximately 5 years. Participants will make multiple visits to the clinic (with some visits optionally conducted by home health) and will have a follow-up assessment 4 weeks after the last dose of study drug.

ELIGIBILITY:
Inclusion criteria:

1. Participant with a diagnosis of NT1 who has completed a controlled study with TAK-861, and for whom the investigator has no clinical objection to their enrollment.

Exclusion criteria:

1. Participant has a treatment-emergent adverse event (TEAE) that remains severe at the time of rollover related to the study drug from the parent study or discontinued because of TEAEs in the parent study.
2. Participant has a risk of suicide according to endorsement of item 4 or 5 on the Columbia Suicide Severity Rating Scale (C-SSRS).
3. The participant has alanine aminotransferase (ALT) or aspartate aminotransferase (AST) values >1.5 times the upper limit of normal (ULN).
4. Participant has a current medical disorder, other than narcolepsy with or without cataplexy, associated with excessive daytime sleepiness (EDS).
5. Participant has current active major depressive episode (MDE) or has had an active MDE in the past 6 months.
6. Participant has developed (within the last 6 months) gastrointestinal disease that is expected to influence the absorption of drugs.
7. Participant has epilepsy or history of seizure.
8. Participant has any other medical condition, such as anxiety, depression, heart disease, or significant hepatic, pulmonary, or renal disease, that requires them to take excluded medications.
9. Participant has a history of cerebral ischemia, transient ischemic attack (<5 years ago), or cerebral hemorrhage.
10. Participant has a history of myocardial infarction, clinically significant coronary artery disease, clinically significant angina, clinically significant cardiac rhythm abnormality, or heart failure.
11. Participant has a history of cancer in the past 5 years.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-04-05 (Actual); Primary Completion 2028-02-28 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With at Least One or More Treatment-emergent Adverse Events (TEAEs) | From signing the informed consent form up to follow-up of 4 weeks after the last dose (Up to approximately 5 years)
  An adverse event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (e.g., a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A TEAE is defined as an adverse event with an onset that occurs after receiving study drug.

SECONDARY OUTCOMES:
Change from Baseline in the Parent Study in Mean Sleep Latency from the Maintenance of Wakefulness Test (MWT) | Baseline (parent study), Week 26 (current LTE study)
  The MWT evaluates a person's ability to remain awake under soporific conditions. Because there is no biological measure of wakefulness, wakefulness is measured indirectly by the tendency to fall asleep. This tendency to fall asleep is measured via electroencephalography-derived sleep latency in the MWT. The MWT consists of four 40-minute sessions done 2 hours apart. Sleep latency in each session will be recorded. Participants will be required to stay awake in between the 4 sessions.
Change from Baseline in the Parent Study in Epworth Sleepiness Scale (ESS) Total Score | Baseline (parent study); Week 2 through Year 5 (current LTE study)
  The ESS provides individuals with 8 different situations of daily life and asks them how likely they are to fall asleep in those situations (scored 0 to 3) and to try to imagine their likelihood of dozing even if they have not actually been in the identical situation; the scores are summed to give an overall score of 0 to 24. Higher scores indicate stronger subjective daytime sleepiness, and scores below 10 are considered to be within the normal range.
Change from Baseline in the Parent Study in Weekly Cataplexy Rate (WCR) Using the Patient-reported Cataplexy Diary | Baseline (parent study); Year 1 through Year 5 (current LTE study)
  Participants will record episodes of cataplexy in the diary throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (52):
- United States (19):
  - Sleep Disorders Center of Alabama, Birmingham, Alabama
  - Stanford Center for Sleep Sciences and Medicine, Redwood City, California
  - SDS Clinical Trials, Inc., Santa Ana, California
  - Delta Waves LLC - Hunt - PPDS, Colorado Springs, Colorado
  - Florida Pediatric Research Institute, Orlando, Florida
  - Neurotrials Research, Atlanta, Georgia
  - Georgia Neuro Center, Gainesville, Georgia
  - Neurocare Inc, Newton, Massachusetts
  - Henry Ford Medical Center - Columbus, Novi, Michigan
  - Research Carolina Elite, Denver, North Carolina
  - ARSM Research, LLC, Huntersville, North Carolina
  - CTI Research Center, Cincinnati, Ohio
  - Intrepid Research, Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio Sleep Medicine Institute, Dublin, Ohio
  - Medical University of South Carolina - PPDS, Charleston, South Carolina
  - Bogan Sleep Consultants, LLC, Columbia, South Carolina
  - Sleep Therapy and Research Center, San Antonio, Texas
  - Children's Specialty Group, Norfolk, Virginia
- Woolcock Institute of Medical Research, Glebe, New South Wales, Australia
- Terveystalo Helsinki Sleep Clinic, Helsinki, Uusimaa, Finland
- France (4):
  - Hopital Pierre-Paul Riquet, Toulouse, Haute-Garonne
  - CHU Gui De Chauliac, Montpellier, Herault
  - CHU de Grenoble, La Tronche, Isere
  - Hopital de la Pitie Salpetriere, Paris
- Germany (4):
  - Universitaet Regensburg am Bezirksklinikum, Regensburg, Bavaria
  - Somni Bene Institut fur Medizinische Forschung und Schlafmedizin Schwerin GmbH, Schwerin, Mecklenburg-Vorpommern
  - Charite - Universitatsmedizin Berlin, Berlin
  - Klinische Forschung Hamburg, Hamburg
- Italy (3):
  - Fondazione PTV Policlinico Tor Vergata, Rome, Lazio
  - Istituto Neurologico Mediterraneo Neuromed, Pozzilli, Molise
  - Ospedale Bellaria, Bellaria
- Japan (6):
  - Kurume University Hospital, Kurume-Shi, Hukuoka
  - Howakai Kuwamizu Hospital, Kumamoto, Kumamoto
  - YOU ARIYOSHI Sleep Clinic, Nagasaki, Nagasaki
  - Gokeikai Osaka Kaisei Hospital, Osaka, Osaka
  - Koishikawa Tokyo Hospital, Bunkyo-Ku, Tokyo
  - Aichi Medical University Hospital, Nagakute
- Netherlands (2):
  - Kempenhaeghe - PPDS, Heeze, North Brabant
  - Slaap-Waakcentrum SEIN Heemstede, Heemstede, North Holland
- University of Oslo, Oslo, Norway
- Spain (7):
  - Hospital Universitario Araba Santiago, Vitoria-Gasteiz, Alava
  - Hospital General de Castello, Castellon, Castellon
  - Hospital de La Ribera, Alzira, Valencia
  - Hospital Universitario Vall d'Hebron - PPDS, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Instituto de Investigaciones del Sueno, Madrid
  - Hospital Vithas Madrid Arturo Soria, Madrid
- Sahlgrenska University Hospital, Gothenburg, Västra Götaland County, Sweden
- Switzerland (3):
  - Klinik Barmelweid AG, Barmelweid, Aargau (de)
  - Neurocenter of Southern Switzerland, Lugano, Ticino (it)
  - Universitaetsspital Bern - Inselspital, Bern

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link. — https://clinicaltrials.takeda.com/study-detail/5daa86dd644c4a8c?idFilter=%5B%22TAK-861-2003%22%5D